CLINICAL TRIAL: NCT05664997
Title: Relationship Between Playing-Related Factors and Occupational Balance in Professional Violinists
Brief Title: Playing-Related Factors and Occupational Balance
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hulya Yucel, Assoc. Prof., Saglik Bilimleri Universitesi
Other Study IDs: 22/286-14/03
Record Dates: First submitted 2022-11-30; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Occupational Balance; Posture
Keywords: Functionality; Playing-related pain; Posture; Occupational balance; Violinists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- violinists: musicians who play the violin in a conservatory or orchestra
  Interventions: Behavioral: playing assessment

INTERVENTIONS:
Behavioral: playing assessment — Investigators used Edinburgh Handedness Inventory, the Wong-Baker Faces Pain Rating Scale, the Disability of Arm, Shoulder and Hand - Sports/Musicians (DASH-SM), the Rapid Upper Limb Assessment, and the 11-item revised version of the Occupational Balance Questionnaire (OBQ11 - T). All have their Turkish validity studies. A correlation analysis was performed to examine the relationship between the variables.

SUMMARY:
As the violin is the riskiest string instrument played by Turkish musicians, violinists were chosen for the sample in this study. The aim of this study was to investigate the relationship between posture, pain, functionality and occupational balance in violinists. The hypothesis was that good playing posture, lack of pain, and functionality affect occupational balance positively.

DETAILED DESCRIPTION:
Occupational balance is the participation in and satisfaction derived from different elements of daily life, including work. Playing performance affects occupational balance of musicians so that complaints arising from the playing of their instruments may negatively affect occupational balance. Forty-five violinists at six different symphony orchestras and conservatories in Istanbul were included. The Personal Information Form, the Edinburgh Handedness Inventory, the Wong-Baker Faces Pain Rating Scale, the Disability of Arm, Shoulder and Hand - Sports/Musicians (DASH-SM), the Rapid Upper Limb Assessment, and the 11-item revised version of the Occupational Balance Questionnaire (OBQ11 - T) were used. Spearman correlation analysis was performed to examine the relationship between the variables.

ELIGIBILITY:
Inclusion Criteria:

* to play the violin in a conservatory or orchestra,
* to be at least 18 years old,
* to volunteer to participate in this study.

Exclusion Criteria:

* Those who played any other instrument professionally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: violinists at Cemal Resit Rey Symphony Orchestra, Maltepe University Conservatory, Istanbul University State Conservatory, Okan University Conservatory, Cemal Resit Rey Jazz Orchestra and Cemal Resit Rey Youth Orchestra.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
occupational balances of the violinists | 25 minutes
  Occupational balances of the violinists change with playing posture, pain, and functionality of upper extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Yucel, Assoc. Prof., Study Chair — Saglik Bilimleri University
Locations (1):
- Hulya Yucel, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Musicians' medicine: musculoskeletal problems in string players. — https://pubmed.ncbi.nlm.nih.gov/24009899/
- See also: Occupational balance as used in occupational therapy: a concept analysis. — https://pubmed.ncbi.nlm.nih.gov/21780985/
- See also: Comparing violinists' body movements while standing, sitting, and in sitting orientations to the right or left of a music stand. — https://pubmed.ncbi.nlm.nih.gov/24925176/